CLINICAL TRIAL: NCT02266797
Title: Effect of Intravenous Corticosteroid Injections on Dysphagia After Anterior Cervical Spine Surgery: a Randomized, Double-blind, Placebo-controlled Study
Brief Title: Effect of Intravenous Corticosteroid Injections on Dysphagia After Cervical Spine Surgery
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13-00108
Record Dates: First submitted 2014-10-02; First posted 2014-10-17 (Estimated); Results first posted 2016-03-14 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-09

CONDITIONS: Dysphagia After Anterior Cervical Decompression and Fusion of the Spine
MeSH Terms: interventions — Dexamethasone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexamethasone (Active Comparator): Subject will receive doses of intravenous dexamethasone, a corticosteroid. The first dose will be given before the incision and the subsequent doses will be given 8 and 16 hours after the first dose. Dexamethasone doses will be 0.3 mg/kg for the first dose and 0.15 mg/kg for each subsequent dose.
  Interventions: Drug: Dexamethasone
- Saline (Placebo Comparator): Subject will receive doses of intravenous physiological saline solution.
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Dexamethasone — The first dose will be given before the incision and the subsequent doses will be given 8 and 16 hours after the first dose. Dexamethasone doses will be 0.3 mg/kg for the first dose and 0.15 mg/kg for each subsequent dose.
  Arms: Dexamethasone
Other: Saline — The first dose will be given before the incision and the subsequent doses will be given 8 and 16 hours after the first dose.
  Arms: Saline

SUMMARY:
This is a randomized, double-blind, placebo-controlled study to examine the effect of local intravenous steroids following anterior cervical spine surgery on the development of dysphagia in patients.

DETAILED DESCRIPTION:
The purpose of this randomized, double-blind, placebo-controlled study is to examine the effect of local intravenous steroids following anterior cervical spine surgery on the development of dysphagia in patients. This study aims to investigate if there is a difference in the efficacy of intravenous steroids compared to a placebo of physiological saline for patients undergoing anterior cervical spine surgery. Furthermore, this study aims to investigate the correlation between radiographic measurements of soft tissue swelling and the severity of dysphagia for patients. Finally, this study aims to examine the impact of intravenous steroids on nausea and radicular pain in patients. Secondary outcome measures will include patient focused outcomes questionnaires, pain medication requirements, and fusion rates.

ELIGIBILITY:
Inclusion Criteria:

* The subjects included in the study are patients undergoing an anterior cervical spine procedure.

Exclusion Criteria:

* Patients with greater than ASA grade II will be excluded. Patients with non-degenerative conditions, such as trauma, tumors, infection, radiation, and diabetes will be excluded. Patients with posterior procedures will be excluded. Patients with clinical pre-operative dysphagia, indicated by a score of 3 or higher on the EAT-10 questionnaire,19 will also be excluded. Patients who are pregnant will be excluded from this study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-11; Primary Completion 2015-09-01 (Actual); Study Completion 2015-09-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Center for Musculoskeletal Care (CMC), New York, New York
  - NYU Langone Medical Center, New York, New York
  - NY Spine Institute, Westbury, New York

REFERENCES:
- [Background] Leonard R, Belafsky P. Dysphagia following cervical spine surgery with anterior instrumentation: evidence from fluoroscopic swallow studies. Spine (Phila Pa 1976). 2011 Dec 1;36(25):2217-23. doi: 10.1097/BRS.0b013e318205a1a7. PMID 21325988
- [Background] Bazaz R, Lee MJ, Yoo JU. Incidence of dysphagia after anterior cervical spine surgery: a prospective study. Spine (Phila Pa 1976). 2002 Nov 15;27(22):2453-8. doi: 10.1097/00007632-200211150-00007. PMID 12435974
- [Background] Stewart M, Johnston RA, Stewart I, Wilson JA. Swallowing performance following anterior cervical spine surgery. Br J Neurosurg. 1995;9(5):605-9. doi: 10.1080/02688699550040882. PMID 8561932
- [Background] Winslow CP, Winslow TJ, Wax MK. Dysphonia and dysphagia following the anterior approach to the cervical spine. Arch Otolaryngol Head Neck Surg. 2001 Jan;127(1):51-5. doi: 10.1001/archotol.127.1.51. PMID 11177014
- [Background] Martin RE, Neary MA, Diamant NE. Dysphagia following anterior cervical spine surgery. Dysphagia. 1997 Winter;12(1):2-8; discussion 9-10. doi: 10.1007/pl00009513. PMID 8997826

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexamethasone | Saline
Started | 1 | 3
Completed | 1 | 2
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone | Saline | Total
Number analyzed (Participants) | 1 | 3 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 4
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Intravenous Corticosteroids Effect on Post-operative Dysphagia
Description: The severity of dysphagia will be evaluated by dysphagia questionnaires and a two week postoperative swallow evaluation by a licensed swallowing expert. If recommended by the swallow evaluation, a videofluoroscopic swallow study (VFSS) will be performed to further evaluate the severity of dysphagia.
Time Frame: 12 months
Population: Data not available due to premature halting of study
Arm/Group | Dexamethasone | Saline
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: The Correlation Between Radiographic Data and the Extent of Dysphagia in Patients.
Description: Soft-tissue swelling will be measured by the anterior cervical soft-tissue shadow width on lateral cervical radiographs. The extent of dysphagia will be evaluated by the dysphagia questionnaires, the swallow evaluation, and the VFSS, if necessary.
Time Frame: 12 months
Population: Data not available due to premature halting of study
Arm/Group | Dexamethasone | Saline
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: The Efficacy of Intravenous Steroids on Aspiration Rates of Patients Undergoing Anterior Cervical Spine Surgery.
Description: Aspiration rates will be evaluated by the percentage of patients in each group with post-operative aspiration.
Time Frame: 12 months
Population: Data not available due to premature halting of study
Arm/Group | Dexamethasone | Saline
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Examine the Impact of Dexamethasone on the Development of Postoperative Nausea.
Description: This will be quantified by the visual analogue scale (VAS) questionnaire for nausea and measuring the number of vomiting episodes following surgery.
Time Frame: Immediate post-operatively
Population: Data not available due to premature halting of study
Arm/Group | Dexamethasone | Saline
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Examine the Impact of Dexamethasone on Radicular Pain.
Description: This will be quantified by the NDI questionnaire and VAS questionnaire for neck pain and arm pain.
Time Frame: 12 months
Population: Data not available due to premature halting of study
Arm/Group | Dexamethasone | Saline
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Examine Whether Intravenous Steroids Affect the Outcomes of Surgery, for Example, Fusion Rates.
Description: The outcomes of surgery will be examined through the 1 year post-operative appointment.
Time Frame: 12 months
Population: Data not available due to premature halting of study
Arm/Group | Dexamethasone | Saline
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Dexamethasone | Saline
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/3
Other Adverse Events (participants affected / at risk) | 0/1 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes